CLINICAL TRIAL: NCT02949388
Title: A Randomized, Double Blind, Parallel Group, Placebo-controlled Trial to Study the Efficacy and Safety of Two Oral Doses of Prurisol Administered Twice Daily for Twelve Weeks to Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Prurisol Administered Orally for Active Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovation Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTIX-PRU-005
Record Dates: First submitted 2016-10-14; First posted 2016-10-31 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Chronic Stable Plaque Psoriasis
MeSH Terms: interventions — BID protein, human; abacavir hydroxyacetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Comparator: Placebo daily Two (2) placebo capsules given twice daily (AM and PM) for 84 (± 2 days
  Interventions: Drug: Placebo
- 300 mg (150 mg BID) (Active Comparator): Active Comparator: 300 mg of Prurisol daily One (1) capsule containing 100 mg Prurisol and one (1) capsule containing 50 mg of Prurisol given twice (AM and PM) for 84 (± 2) days
  Interventions: Drug: 300 mg (150 mg BID)
- 400 mg (200 mg BID) (Active Comparator): Active Comparator: 400 mg of Prurisol daily Two (2) capsule each containing 100 mg Prurisol given twice daily (AM and PM) for 84 (± 2) days
  Interventions: Drug: 400 mg (200 mg BID)

INTERVENTIONS:
Drug: Placebo — Two capsules (both containing Placebo enclosed) taken twice a day and approximately 12 hours apart
  Arms: Placebo
Drug: 400 mg (200 mg BID) — Two capsules (both containing two 50mg tablets enclosed) taken twice a day and approximately 12 hours apart
  Other Names: Prurisol
  Arms: 400 mg (200 mg BID)
Drug: 300 mg (150 mg BID) — Two capsules (one containing 50mg tablet and one containing two 50 mg tablets) taken twice a day and approximately 12 hours apart
  Other Names: Prurisol
  Arms: 300 mg (150 mg BID)

SUMMARY:
This study is designed as a randomized, double blind, parallel group, placebo-controlled trial to study the efficacy and safety of two oral doses of Prurisol administered twice daily for twelve weeks to subjects with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
This study is designed as a randomized, double blind, parallel group, placebo-controlled trial to study the efficacy and safety of two oral doses of Prurisol administered twice daily for twelve weeks to subjects with moderate to severe chronic plaque psoriasis.

Approximately 189 study participants will be enrolled. Subjects will be randomly assigned to one of three treatment groups in a 3:3:1 randomization ratio, respectively.

* Group A (n=81): Prurisol 150 mg bid
* Group B (n=81): Placebo
* Group C (n=27): Prurisol 200 mg bid Outpatient subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy will be recruited to the study. Study participants are required to have a Psoriasis Area and Severity Index (PASI) score ≥ 12, body surface area involvement ≥ 10%, and a static Physician's Global Assessment (sPGA) of moderate or severe (score of 3 or 4).

A subject studied under this clinical protocol will commence with a screening period of up to 4 weeks, a treatment period of 12 weeks, and a follow-up period of 4 weeks ending with an End of Study evaluation.

During treatment, subjects will return to the study center every 2 weeks. Efficacy assessments, including physician and patient rated endpoints, will be measured throughout the study. Safety and tolerability will be assessed by ascertainment of AEs and results of clinical laboratory testing, vital signs assessments, and need for concomitant medications.

At a subset of sites, blood samples for determination of plasma concentrations of Prurisol (abacavir glycolate) and abacavir, it's metabolite, will be obtained from subjects who consent to provide these samples. At selected sites, for those subjects consenting to photography, standardized digital photographs will be obtained for illustrative purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated written informed consent to participate in the clinical study
2. Male or non-pregnant female adults at least 18 years of age at time of informed consent
3. Chronic plaque-type psoriasis diagnosed for at least 6 months prior to baseline (at time of first study dose)
4. Moderate to severe plaque psoriasis as defined at baseline by:

   1. PASI score of 12 or greater, and
   2. Static PGA score of moderate (3) or severe (4), and
   3. Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater
5. Candidate for systemic therapy or phototherapy
6. Willing to limit ultraviolet light exposure from sunbathing, use of tanning booths, prolonged outdoor exposure, or from other UV light sources during the study.
7. Willing and able to comply with scheduled visits, study assessments and l laboratory tests, and other study procedures

Exclusion Criteria:

1. Positive blood test for HLA-B*5701 allele
2. Currently have forms of psoriasis other than chronic plaque-type, (e.g., guttate, erythrodermic, exfoliative, palmoplantar, pustular), with the exception of nail psoriasis
3. Evidence of drug-induced psoriasis, e.g., a new onset or current exacerbation of psoriasis from beta-blockers, calcium channel inhibitors, antimalarial drugs or lithium
4. Psoriasis flare or rebound within 4 weeks prior to Screening
5. Active inflammatory diseases other than psoriasis that might confound the evaluation of study treatment on signs and symptoms of psoriasis.
6. . Any of the following prohibited treatments that do not meet the specified minimum washout period:

   1. Biologic immunomodulating treatments of brodalumab or ustekinumab within 24 weeks prior to start of study treatment
   2. Biologic immunomodulating treatments such as adalimumab, etanercept, infliximab, ixekizumab, secukinumab or certolizumab pegol within 12 weeks prior to start of study treatment
   3. Systemic immunomodulating treatments other than biologics within 4 weeks prior to start of study treatment, e.g., oral corticosteroids, injectable corticosteroids (intraarticular, intramuscular, cutaneous/subcutaneous or intravenous), methotrexate, cyclosporine, cyclophosphamide, apremilast

      * Inhaled or intranasal corticosteroids with predominantly local effect (e.g., to treat asthma) are allowable
      * Use of corticosteroids in the eye or the ear are allowable
   4. Other systemic treatments for psoriasis within 4 weeks prior to start of study treatment, e.g., retinoids, fumarates

      * Any such treatment used to treat a symptom of psoriasis but not the condition itself (e.g., anti-histamines for pruritus) is not restricted
   5. Photochemotherapy, e.g., Psoralens + UVA phototherapy (PUVA), within 4 weeks prior to start of study treatment
   6. Phototherapy, e.g., UVA, UVB, within 2 weeks prior to start of study treatment
   7. Topical treatments that could affect signs and symptoms of psoriasis within 2 weeks prior to start of study treatment, e.g., corticosteroids, vitamin D analogs, retinoids, pimecrolimus, tacrolimus, tars, keratolytics

      * Allowable exceptions are: low or least potent (Class 6 or 7) topical corticosteroids for use on face, palms, soles, and intertriginous areas only; tar and salicylic acid preparations/shampoos for use on scalp only; bland emollient for use on any body region
7. Past vaccination with live vaccine within 6 weeks prior to start of study treatment, or plans for administration during the study
8. Any investigational or experimental therapy or procedure or participation in any interventional trial within 4 weeks or 5 half-lives (whichever is longer) prior to start of study treatment
9. Women of child-bearing potential who are not using reliable means of contraception, e.g., abstinence, surgical sterilization (hysterectomy and/or bilateral oophorectomy or partner vasectomy) or tubal ligation, double barrier method, oral/ injected/ implanted/ transdermal hormonal contraception, intrauterine device or intrauterine system, throughout study participation, and for 4 weeks after the end of treatment
10. Women of child-bearing potential who are pregnant or nursing (lactating), or planning a pregnancy while participating in the study
11. History of any ongoing, chronic or recurrent infectious disease (with the exception of episodic herpes labialis and herpes genitalis, and vaginal yeast infections)
12. Evidence of tuberculosis infection as defined by a positive QuantiFERON®-TB Gold In-Tube test (QFT-G) at Screening, or subjects with an indeterminate QFT-G test result with any retest result as indeterminate or positive
13. History of either untreated or incompletely treated latent or active tuberculosis infection
14. Ongoing or recent history of any non-psoriatic uncontrolled (in the Investigator's medical opinion) systemic disease, including, but not limited to renal, hepatic, hematologic, gastrointestinal, endocrine, metabolic, pulmonary, cardiac, neurologic, or psychiatric disease. (e.g., A past or current history of hypertension that is controlled with diet and/or medications is not exclusionary.)
15. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years with the exception of: basal cell or squamous cell carcinoma or actinic keratoses that have been treated or excised with no evidence of recurrence in the past 12 weeks; cervical carcinoma in situ or non-invasive malignant colon polyps that have been removed
16. Active systemic infections during the past two weeks (exception: common cold) prior to start of study treatment or any infection that reoccurs on a regular basis
17. Past medical history of infection with HIV, hepatitis B or hepatitis C
18. History of any allergic reaction to any formulation of abacavir
19. Previous treatment with any abacavir-containing product, e.g., Ziagen®, Epzicom®, or Trizivir®
20. Previous participation in a clinical study of Prurisol
21. Presence of any medical or psychiatric condition that, in the Investgator's opinion, makes it unlikely that the requirements of the protocol will be completed
22. History of alcohol or substance abuse, unless in full remission for more than 6 months prior to start of study treatment
23. Electrocardiogram (ECG) obtained at Screening visit which shows medically relevant abnormalities which may affect subject safety or interpretation of study results
24. Observed clinical laboratory values/abnormalities during Screening that show any one or more of the following:

    1. Screening total white blood cell (WBC) count <2.5 x 10^9/L, or platelets <100 x 10^9/L or neutrophils <1.2 x 10^9/L or hemoglobin <8.5 g/dL
    2. Screening serum creatinine level exceeding 2.0 mg/dL (176.8 µmol/L)
    3. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 2 x ULN
25. Any other severe acute or chronic medical or psychiatric condition or test abnormality(ies) that, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving at least a 75% reduction from baseline in PASI score (PASI75) at Week 12 | 12 Weeks
  The Psoriasis Area and Severity Index (PASI) quantifies the severity of psoriasis based on lesion severity and the percent of body surface area affected. It is a composite assessment, across body regions, reflected in a single score: 0 (no disease) to 72 (maximal disease).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 16 Weeks
  Reporting of Adverse Events measurements, and reporting of adverse events.

SECONDARY OUTCOMES:
Proportion of subjects achieving a static Physician Global Assessment (sPGA) score of clear (0) or almost clear (1) with at least a 2-point reduction from baseline | 16 Weeks
  The static Physician Global Assessment reflects an overall severity of the erythema, induration and scaling across all psoriatic lesions on a 5-point scale, where 0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe.
PASI75 response at time points through Week 16 | 16 Weeks
  The Psoriasis Area and Severity Index (PASI) quantifies the severity of psoriasis based on lesion severity and the percent of body surface area affected. It is a composite assessment, across body regions, reflected in a single score: 0 (no disease) to 72 (maximal disease).
The actual and change from baseline in patient-reported itch severity score | 16 weeks
  The severity of itching due to psoriasis will be assessed on a horizontal numeric rating scale, anchored by the terms "No itching" (0) and "Worst possible itching" (10).
Assessment of patient-reported quality of life by the Dermatology Life Quality Index (DLQI) | 16 Weeks
  The Dermatology Life Quality Index (DLQI) is a 10-item general dermatology questionnaire that assesses patient health-related quality of life in adult subjects with skin diseases such as psoriasis
Assessment of patient-reported quality of life by the Short Form-36 Health Survey (version 2, acute form) | 12 Weeks
  The SF-36 is a widely used general health status questionnaire that assesses 8 domains of functional health and well-being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions
Assessment of patient-reported quality of life by the Euro-Qol 5 Dimensions Health State Profile | 12 Weeks
  The EQ-5D is a generic instrument designed to assess a subject's general health status. The instrument consists of a questionnaire and a visual analog scale (VAS)
Assessment of Patient Satisfaction with Study Treatment (PSST) | 12 Weeks
  Overall patient satisfaction with study treatment will be assessed on a 7-point rating scale, with response options range from "very dissatisfied" to "very satisfied"
Plasma concentrations of Prurisol | 4 Weeks
  Measurement of Prurisol (abacavir glycolate) from a subset of subjects in the trial
Plasma concentrations of abacavir | Timeframe: 4 weeks
  Measurement of abacavir, a metabolite of Prurisol, from a subset of subjects in the trial

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Study Site, Glendale, Arizona
  - Study Center, Hot Springs, Arkansas
  - Clinical Study Site, Rogers, Arkansas
  - Study Center, Los Angeles, California
  - Study Site, Los Angeles, California
  - Clinical Study Site, Murrieta, California
  - Clinical Study Site, Oceanside, California
  - Study Site, Sherman Oaks, California
  - Study Site, Denver, Colorado
  - Clinical Study Site, Denver, Colorado
  - Study Site, Port Orange, Florida
  - Clinical Study Site, Tampa, Florida
  - Study Site, Savannah, Georgia
  - Study Center, Arlington Heights, Illinois
  - Clinical Study Site, South Bend, Indiana
  - Study Center, Overland Park, Kansas
  - Study Site, Louisville, Kentucky
  - Clinical Study Site, Clarkston, Michigan
  - Clinical Study Site, Clinton Township, Michigan
  - Clinical Study Site, St Louis, Missouri
  - Study Site, Las Vegas, Nevada
  - Clinical Study Site, Portsmouth, New Hampshire
  - Clinical Study Site, Berlin, New Jersey
  - Clinical Study Site, New York, New York
  - Clinical Study Site, Portland, Oregon
  - Study Site, Johnston, Rhode Island
  - Study Center, Austin, Texas
  - Clinical Study Site, Houston, Texas
  - Clinical Study Site, Pflugerville, Texas
  - Clinical Study Site, San Antonio, Texas
  - Study Site, San Antonio, Texas
  - Study Site, Webster, Texas
  - Study Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No